CLINICAL TRIAL: NCT01273870
Title: Post Marketing Surveillance Investigating Blood Compatibility Characteristics of Baxter Xenium+, Fresenius FX and Gambro Polyflux Dialyzers
Brief Title: Blood Compatibility Characteristics of Baxter Xenium+, Fresenius FX and Gambro Polyflux Dialyzers
Status: Completed | Type: Observational
Sponsor: Praxisverbund Dialyse und Apherese (Other)
Responsible Party: Dr. Peter Ahrenholz, BioArtProducts GmbH, Rostock, Germany
Other Study IDs: PDA-02
Record Dates: First submitted 2010-12-22; First posted 2011-01-11 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2010-11

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: hemodialysis; high-flux-dialyzer; performance; blood compatibility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the dialyzer evaluation is to compare performance characteristics and haemocompatibility of the Baxter Xenium+ (Polynephron), Fresenius FX and Gambro Polyflux dialyzers

DETAILED DESCRIPTION:
The Xenium+ is a new high flux dialyzer made from Polynephron membrane designed and manufactured by the Nipro Company in Japan. This dialyzer has been subjected to in-vitro testing, and all legally required biological safety tests have been conducted and CE-mark was granted in June 2010. Xenium+ has the same Polynephron membrane as the Xenium family of dialyzers which has been available commercially globally for approximately three years. Clinical evaluations have been completed with the Polynephron membrane within the last three years. The improvement in the Xenium+ line is that the casing is now made from polypropylene.

The aim of the dialyzer evaluation is to compare performance characteristics and hemocompatibility of the Xenium+ (Polynephron), Fresenius FX and Gambro Polyflux dialyzers.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients 18 years or older
* Stable on hemodialysis for more than 3 months
* An average haematocrit value of 30 % or higher in the last three 3 months
* Stable vascular access of either a fistula or graft
* Stable anticoagulation and regimen
* Stable erythropoiesis-stimulating agent (ESA) regimen for the last three 3 months
* No active infection
* Able to sign informed consent and able to participate in the study
* Medically stable

Exclusion Criteria:

* Participation in another study which may interfere with the planned study
* Active infection
* Medical conditions which may interfere with the study (cardiac, liver disease, hepatitis)
* Female(s) who are pregnant or planning to be pregnant
* Problem with or allergy to anticoagulation
* Central venous catheters

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 8 patients will undergo 1 treatment each with the 4 high-flux dialyzer types using a bloodflow of 300 ml/min, dialysate flow 500 ml/min and the dialysis machine Fresenius 5008
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Clearance for urea, phosphate, beta-2-microglobulin blood cell drop, complement factor C5a, TAT | January 2011

SECONDARY OUTCOMES:
General survey of the dialysis treatments | January 2011
  Registration of adverse effects of the dialysis treatments

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Winkler, PhD, Study Director — Praxisverbund fuer Dialyse und Apherese Rostock